CLINICAL TRIAL: NCT03494894
Title: Bacteriological Link Between Upper and Lower Airways in Cystic Fibrosis and Primary Ciliary Dyskinesia
Acronym: BAVASI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: BAVASI
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-07

CONDITIONS: Cystic Fibrosis; Primary Ciliary Dyskinesia
MeSH Terms: conditions — Cystic Fibrosis; Ciliary Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with Cystic Fibrosis and Primary Ciliary Dyskinesia
  Interventions: Diagnostic Test: Middle meatus aspirations and sputum

INTERVENTIONS:
Diagnostic Test: Middle meatus aspirations and sputum — Bacterial genotype sequencing analysis will be performed in patients with bacteriological concordance between upper and lower airways.

SUMMARY:
Cytobacteriological examination of sputum and bacteriological sampling in the middle meatus.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 6 years old
* Patients with cystic fibrosis or primary ciliary dyskinesia.
* Patients capable of performing an expectorations
* Patients having been informed of the research, having received the information note and not having opposed the research

Exclusion Criteria:

- Refusal to participate in the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The protocol will be proposed to the patients followed in the CHI creteil with cystic fibrosis and primary ciliary dyskinesia. Patients should be followed by a lung specialist and ENT specialist and follow the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Presence of bacterial colonization of the upper and lower airway | 1 day

SECONDARY OUTCOMES:
bacteriological concordance | 1 day
  bacteriological concordance of upper airways (VAS) and lower (VAI) between patients with cystic fibrosis and those with primary ciliary dyskinesia.
bacteria genotype | 1 day
  Compare the genotype of bacteria present in both VAS and VAI.
bacteriological concordance in children | 1 day
  Subgroup analysis (group <18 years old)
bacteriological concordance in adult | 1 day
  Subgroup analysis (adult group)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal de Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kahl BC, Duebbers A, Lubritz G, Haeberle J, Koch HG, Ritzerfeld B, Reilly M, Harms E, Proctor RA, Herrmann M, Peters G. Population dynamics of persistent Staphylococcus aureus isolated from the airways of cystic fibrosis patients during a 6-year prospective study. J Clin Microbiol. 2003 Sep;41(9):4424-7. doi: 10.1128/JCM.41.9.4424-4427.2003. PMID 12958283
- [Background] Frederiksen B, Lanng S, Koch C, Hoiby N. Improved survival in the Danish center-treated cystic fibrosis patients: results of aggressive treatment. Pediatr Pulmonol. 1996 Mar;21(3):153-8. doi: 10.1002/(SICI)1099-0496(199603)21:33.0.CO;2-R. PMID 8860069
- [Background] Berkhout MC, van Rooden CJ, Rijntjes E, Fokkens WJ, el Bouazzaoui LH, Heijerman HG. Sinonasal manifestations of cystic fibrosis: a correlation between genotype and phenotype? J Cyst Fibros. 2014 Jul;13(4):442-8. doi: 10.1016/j.jcf.2013.10.011. Epub 2013 Nov 5. PMID 24210900
- [Background] Berkhout MC, Klerx-Melis F, Fokkens WJ, Nuijsink M, van Aalderen WM, Heijerman HG. CT-abnormalities, bacteriology and symptoms of sinonasal disease in children with Cystic Fibrosis. J Cyst Fibros. 2016 Nov;15(6):816-824. doi: 10.1016/j.jcf.2016.03.004. Epub 2016 Apr 3. PMID 27049043
- [Background] Jelsbak L, Johansen HK, Frost AL, Thogersen R, Thomsen LE, Ciofu O, Yang L, Haagensen JA, Hoiby N, Molin S. Molecular epidemiology and dynamics of Pseudomonas aeruginosa populations in lungs of cystic fibrosis patients. Infect Immun. 2007 May;75(5):2214-24. doi: 10.1128/IAI.01282-06. Epub 2007 Jan 29. PMID 17261614
- [Background] Mainz JG, Naehrlich L, Schien M, Kading M, Schiller I, Mayr S, Schneider G, Wiedemann B, Wiehlmann L, Cramer N, Pfister W, Kahl BC, Beck JF, Tummler B. Concordant genotype of upper and lower airways P aeruginosa and S aureus isolates in cystic fibrosis. Thorax. 2009 Jun;64(6):535-40. doi: 10.1136/thx.2008.104711. Epub 2009 Mar 11. PMID 19282318
- [Background] Berkhout MC, Rijntjes E, El Bouazzaoui LH, Fokkens WJ, Brimicombe RW, Heijerman HG. Importance of bacteriology in upper airways of patients with Cystic Fibrosis. J Cyst Fibros. 2013 Sep;12(5):525-9. doi: 10.1016/j.jcf.2013.01.002. Epub 2013 Jan 26. PMID 23357546
- [Background] Aanaes K, Johansen HK, Poulsen SS, Pressler T, Buchwald C, Hoiby N. Secretory IgA as a diagnostic tool for Pseudomonas aeruginosa respiratory colonization. J Cyst Fibros. 2013 Jan;12(1):81-7. doi: 10.1016/j.jcf.2012.07.001. Epub 2012 Jul 20. PMID 22819141
- [Background] Fischer N, Hentschel J, Markert UR, Keller PM, Pletz MW, Mainz JG. Non-invasive assessment of upper and lower airway infection and inflammation in CF patients. Pediatr Pulmonol. 2014 Nov;49(11):1065-75. doi: 10.1002/ppul.22982. Epub 2014 Jan 25. PMID 24464968
- [Background] Aanaes K. Bacterial sinusitis can be a focus for initial lung colonisation and chronic lung infection in patients with cystic fibrosis. J Cyst Fibros. 2013 Sep;12 Suppl 2:S1-20. doi: 10.1016/S1569-1993(13)00150-1. PMID 24064077
- [Background] Magnin ML, Cros P, Beydon N, Mahloul M, Tamalet A, Escudier E, Clement A, Le Pointe HD, Blanchon S. Longitudinal lung function and structural changes in children with primary ciliary dyskinesia. Pediatr Pulmonol. 2012 Aug;47(8):816-25. doi: 10.1002/ppul.22577. Epub 2012 May 8. PMID 22570319
- [Background] Alanin MC, Nielsen KG, von Buchwald C, Skov M, Aanaes K, Hoiby N, Johansen HK. A longitudinal study of lung bacterial pathogens in patients with primary ciliary dyskinesia. Clin Microbiol Infect. 2015 Dec;21(12):1093.e1-7. doi: 10.1016/j.cmi.2015.08.020. Epub 2015 Sep 2. PMID 26341913
- [Background] Alanin MC, Johansen HK, Aanaes K, Hoiby N, Pressler T, Skov M, Nielsen KG, von Buchwald C. Simultaneous sinus and lung infections in patients with primary ciliary dyskinesia. Acta Otolaryngol. 2015 Jan;135(1):58-63. doi: 10.3109/00016489.2014.962185. Epub 2014 Nov 5. PMID 25370419